CLINICAL TRIAL: NCT06863935
Title: A Pilot Study of High-Dose Omega-3 (Soloways ™) Polyunsaturated Fatty Acids in Patients with Dyslipidemia Carrying FADS1/FADS2 Variants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SW021
Record Dates: First submitted 2025-02-20; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Dyslipidemia
Keywords: Genetics; supplements; Omega3; FADS1/FADS2 gene; cholesterol
MeSH Terms: conditions — Dyslipidemias; Pena Shokeir syndrome, type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FADS Variant (Homozygous or High-Risk) Cohort (Experimental)
  Interventions: Dietary Supplement: High-dose omega-3 PUFA supplementation
- Non-Variant (Control) Cohort (Active Comparator)
  Interventions: Dietary Supplement: High-dose omega-3 PUFA supplementation

INTERVENTIONS:
Dietary Supplement: High-dose omega-3 PUFA supplementation — High-dose omega-3 PUFA supplementation (2-4 g/day EPA+DHA) for 12 weeks in addition to standard lipid-lowering therapy
  Arms: FADS Variant (Homozygous or High-Risk) Cohort
Dietary Supplement: High-dose omega-3 PUFA supplementation — High-dose omega-3 PUFA supplementation (2-4 g/day EPA+DHA) for 12 weeks in addition to standard lipid-lowering therapy
  Arms: Non-Variant (Control) Cohort

SUMMARY:
This pilot, genotype-stratified clinical trial aims to evaluate the safety and preliminary efficacy of high-dose omega-3 PUFA supplementation in patients with dyslipidemia who carry a specific "unfavorable" genetic variant in the FADS1/FADS2 gene cluster. The study will compare lipid profile improvements and inflammatory markers between two cohorts: (1) homozygous (or high- risk) carriers of the FADS1/FADS2 variants and (2) non-carriers (wild-type). Investigators hypothesize that individuals with these variants will show a more pronounced reduction in triglyceride levels and inflammatory markers following high-dose omega-3 supplementation due to their diminished endogenous synthesis of long-chain PUFAs.

DETAILED DESCRIPTION:
Dyslipidemia is a key risk factor for cardiovascular disease, often characterized by elevated triglycerides, low HDL cholesterol, and/or high LDL cholesterol. Genetic variants in the fatty acid desaturase genes FADS1 and FADS2 can alter the conversion of shorter-chain polyunsaturated fatty acids into longer-chain forms (EPA, DHA), leading to suboptimal endogenous production of these beneficial fatty acids. Omega-3 supplements, especially EPA and DHA, have been shown to lower triglycerides and modulate inflammatory pathways. This study examines whether high-dose omega-3 supplementation (2-4 g/day) confers greater benefit for carriers of certain "unfavorable" FADS1/ FADS2 polymorphisms, potentially optimizing cardiovascular risk reduction in this genetically defined subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years with documented dyslipidemia (elevated triglycerides and/or LDL cholesterol).

  * On stable lipid-lowering therapy (e.g., statins) or lifestyle regimen for at least 4 weeks prior to enrollment, if applicable.
  * Willingness to undergo genetic testing for FADS1/FADS2 variants. For the FADS Variant Cohort: confirmed homozygous (or high-risk) polymorphisms in FADS1/FADS2.
  * For the Non-Variant Cohort: confirmed wild-type FADS genotype.

Exclusion Criteria:

* Use of prescription omega-3 products or high-dose fish oil supplements within 4 weeks prior to enrollment.
* Known hypersensitivity to fish or fish oil products. Significant renal or hepatic impairment, uncontrolled thyroid disease, or other comorbidities that may confound results.
* Pregnancy or breastfeeding.
* Inability or unwillingness to comply with study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2025-01-18 (Actual)

PRIMARY OUTCOMES:
Percent Change in Triglyceride Levels | Week 12
Percent Change in LDL and HDL Cholesterol | 12 weeks

SECONDARY OUTCOMES:
Change in Inflammatory Markers hs-CRP mg/l | 12 weeks
Any Adverse Events | 12 weeks
Change in Total Cholesterol mmol/l | 12 weeks
Change in Non-HDL Cholesterol mmol/l | 12 weeks
Percent Change in Body Weight | 12 weeks
Change in BMI | 12 weeks
Change in Patient-Reported Quality of Life as Measured by the World Health Organization | 12 weeks
  Patient-reported quality of life will be assessed using the World Health Organization Quality of Life Instrument, Short Form (WHOQOL-BREF). This validated questionnaire provides scores ranging from 0 to 100 for each domain (physical health, psychological health, social relationships, and environment), where higher scores indicate a better quality of life. The outcome will be reported as the mean change in the relevant domain scores from baseline to 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for New Medical Techologies, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No